CLINICAL TRIAL: NCT00357279
Title: A Multi-Center, Double-Blind, Placebo-Controlled Randomized, Efficacy and Safety Study of Denufosol Tetrasodium (INS37217) Inhalation Solution in Patients With Mild Cystic Fibrosis Lung Disease
Brief Title: Study of Denufosol Inhalation Solution in Patients With Mild Cystic Fibrosis Lung Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-108
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — denufosol tetrasodium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo - 0.9% w/v sodium chloride solution
- 2 (Experimental)
  Interventions: Drug: denufosol tetrasodium (INS37217) Inhalation Solution

INTERVENTIONS:
Drug: denufosol tetrasodium (INS37217) Inhalation Solution — Denufosol 60 mg is administered as an inhalation solution, three times daily for six months during the double-blind portion of the study. Subsequently, denufosol 60 mg is administered for an additional six months during the open label safety extension.
  Arms: 2
Drug: Placebo - 0.9% w/v sodium chloride solution — 4.2 mL of solution, allowing delivery of approximately 4 mL into the nebulizer cup for nebulization, three times daily for six months.
  Arms: 1

SUMMARY:
The purpose of this trial is to evaluate the safety and effectiveness of a one dose strength of denufosol compared to placebo in patients with mild CF lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed diagnosis of cystic fibrosis
* Have FEV1 of greater than or equal to 75% of predicted normal for age, gender, and height
* Be able to reproducibly perform spirometry maneuvers
* Be clinically stable for at least 4 weeks prior to screening

Exclusion Criteria:

* Have abnormal renal or liver function
* Have chest x-ray at screening suggesting clinically significant active pulmonary disease
* Be colonized with Burkholderia cepacia
* Have had a lung transplant

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in lung function | 48 weeks

SECONDARY OUTCOMES:
Pulmonary exacerbation | 48 weeks
Requirements for concomitant CF medications | 48 weeks
Quality of Life | 48 weeks

REFERENCES:
- [Derived] Accurso FJ, Moss RB, Wilmott RW, Anbar RD, Schaberg AE, Durham TA, Ramsey BW; TIGER-1 Investigator Study Group. Denufosol tetrasodium in patients with cystic fibrosis and normal to mildly impaired lung function. Am J Respir Crit Care Med. 2011 Mar 1;183(5):627-34. doi: 10.1164/rccm.201008-1267OC. Epub 2010 Dec 17. PMID 21169471